CLINICAL TRIAL: NCT01048060
Title: Consent for Obtaining Additional Bone Marrow Specimens at the Time of a Diagnostic Bone Marrow Procedure
Brief Title: Consent for Obtaining Additional Bone Marrow Specimens at Time of Diagnostic Bone Marrow Procedure
Status: Terminated | Type: Observational
Why Stopped: Business Decision
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: BANKPEDSBMS0001; 78014; SU-11022007-789 (Other: Stanford University)
Record Dates: First submitted 2010-01-11; First posted 2010-01-13 (Estimated); Last update posted 2019-02-11 (Actual); Status verified 2019-02

CONDITIONS: Brain Cancer; Cancer
MeSH Terms: conditions — Brain Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — bone marow

INTERVENTIONS:
Procedure: Bone marrow specimen banking

SUMMARY:
The purpose of this study is to collect bone marrow samples for experimental studies.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are having a bone marrow procedure done as part of their standard oncology work-up will be eligible to be consent on this study.

Exclusion Criteria:

* None.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Subjects who are having a bone marrow procedure done as part of their standard oncology work-up will be eligible to be consent on this study.
Sampling Method: Non-Probability Sample
Enrollment: 334 (Actual)
Dates: Start 2002-02; Primary Completion 2015-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Cancer Research in Future | 1 time
  No new information will be gained form this study. However, the specimens obtained me be used for other studies to progress cancer research in the future.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Neyssa Marina, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States